CLINICAL TRIAL: NCT04980833
Title: A Phase II Study to Evaluate the Long-term Safety and Efficacy of Alpelisib in Patients With PIK3CA-Related Overgrowth Spectrum (PROS) Who Previously Participated in Study CBYL719F12002 (EPIK-P1)
Brief Title: Study Assessing Long-term Safety and Efficacy of Alpelisib in Patients With PIK3CA-Related Overgrowth Spectrum (PROS) Who Previously Participated in Study CBYL719F12002 (EPIK-P1)
Acronym: EPIK-P3
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBYL719F12401; 2023-508522-95-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2021-07-19; First posted 2021-07-28 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: PIK3CA-related Overgrowth Spectrum (PROS)
Keywords: PIK3CA-related overgrowth spectrum (PROS); Alpelisib; BYL719; Adult; Pediatric; Phase II
MeSH Terms: interventions — Alpelisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Alpelisib (Experimental): All participants will receive alpelisib once a day
  Interventions: Drug: Alpelisib

INTERVENTIONS:
Drug: Alpelisib — Participant's treatment plan has been established by the treating physician, within the global compassionate use framework. Doses permitted are 50, 125, 200 and 250 mg.
  Other Names: BYL719

SUMMARY:
This is a prospective interventional Phase II multi center study, open label, preceded by a retrospective non-interventional period, to assess the long-term safety and efficacy of alpelisib, in pediatric and adult participants with PROS.

DETAILED DESCRIPTION:
The study will enroll males and females aged ≥2 years who previously participated in EPIK-P1 study and who continued to receive treatment with alpelisib after the cut-off date used in EPIK-P1 (NCT04285723).

The study has an initial retrospective period and a subsequent prospective period.

The retrospective period, is a non-interventional study period and will start one day after the EPIK-P1 data cut-off date (i.e. 10-Mar-2020). It will end the day before the first interventional dose of alpelisib is administered in the prospective period of this study (Day -1). Key safety and efficacy information that was previously collected as per local medical practice and recorded in the medical charts of eligible participants will be longitudinally abstracted.

The prospective period, is an interventional study period and will start on the day of the first interventional dose administration in the prospective period. It will end after all participants have completed at least 5 years of treatment in the prospective period of the study or discontinued earlier, whichever occurs earlier. During this study period, safety and efficacy data will be prospectively collected following a structured plan that is common to all participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants who had previously participated in the study EPIK-P1.
* Signed informed consent form and assent (when applicable) from the participant, parent, or guardian must be obtained prior to any study related screening procedures being performed.
* Participant is treated with at least one dose of alpelisib after the EPIK-P1 study data cut- off date of 09-Mar-2020.

Exclusion Criteria:

For participants in the retrospective period

- All EPIK-P1 participants who permanently discontinued the investigational drug on or prior to the cut-off date 09-Mar-2020.

For participants in the prospective period

* Previous alpelisib treatment discontinuation (after 09-Mar-2020) due to any of the following adverse events:

  * Grade 4 skin and subcutaneous tissue disorders
  * Stevens-Johnson-Syndrome (SJS)/ Toxic Epidermal Necrolysis (TEN) or other SJS/TEN-like severe skin reactions (any grade)
  * Grade 4 hyperglycemia without confounding factors
  * Pneumonitis (any grade)
  * Grade 4 stomatitis
  * Grade 4 pancreatitis
  * Recurrent grade 4 thrombocytopenia
  * Grade 3 or 4 serum creatinine increase
  * Grade 4 isolated total bilirubin elevation
  * Recurrent grade 3 or 4 QT interval corrected by Fridericia's formula prolongation (>500 ms or >60 ms change from baseline)
* Known impairment of GI function due to concomitant disease that may significantly alter the absorption of the study drug (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection) at time of informed consent.
* Participant with uncontrolled diabetes mellitus (Type I or II) at time of informed consent.

Other inclusion/exclusion criteria may apply

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2027-07-22 (Estimated); Study Completion 2027-07-22 (Estimated)

PRIMARY OUTCOMES:
Prospective period only: Proportion of participants with new or worsening grade ≥3 treatment emergent adverse events (AEs) | From date of first interventional dose administration in the prospective period (Day 1) to 30 days after last dose of study drug, assessed up to 5 years.
  Incidence of new or worsening grade ≥3 treatment emergent AEs (by system organ class and preferred term)

SECONDARY OUTCOMES:
Retrospective period: Proportion of participants with Adverse Events (AEs) | From 10-Mar-2020 (1 day after EPIK-P1 data cut-off date) to the day before the first interventional dose of alpelisib is administered in the prospective period of this study (Day -1)
  Incidence, type and severity per common terminology criteria for AEs (CTCAE) v4.03 criteria, causality assessments of AEs, including changes in laboratory values, vital signs and assessment of cardiac function during the retrospective period.
Prospective period: Proportion of participants with AEs | From Day 1 up to 5 years
  Incidence, type and severity per CTCAE v4.03 criteria, causality assessments of AEs, including changes in laboratory values, vital signs, assessment of cardiac function, and growth, sexual maturation and bone/dental development (for applicable age) during the prospective period.
Retrospective and prospective period: Overall clinical assessment as assessed by the investigator | Retrospective: From 10-Mar-2020 (1 day after EPIK-P1 data cut-off date) to the day before the first interventional dose of alpelisib is administered in the prospective period of this study (Day -1). Prospective: From Day 1 up to 5 years
  Proportion of participants with overall clinical assessment reported as improvement, stable or worsened, as assessed by the investigator.
Retrospective and prospective period: Incidence of PROS-related symptoms and complications/comorbidities among participants with symptoms and complications/comorbidities. | Retrospective: From 10-Mar-2020 (1 day after EPIK-P1 data cut-off date) to the day before the first interventional dose of alpelisib is administered in the prospective period of this study (Day -1). Prospective: From Day 1 up to 5 years
  Incidence of symptoms and complications/comorbidities (including taken treatment measures) associated with PROS over time among participants with symptoms and complications/comorbidities.
Retrospective and prospective period: Proportion of participants with healthcare visits/hospitalizations due to PROS. | Retrospective: From 10-Mar-2020 (1 day after EPIK-P1 data cut-off date) to the day before the first interventional dose of alpelisib is administered in the prospective period of this study (Day -1). Prospective: From Day 1 up to 5 years
  Proportion of participants with healthcare visits/hospitalizations due to PROS will be assessed.
Retrospective and prospective period: Proportion of participants requiring PROS-related treatment(s) other than alpelisib | Retrospective: From 10-Mar-2020 (1 day after EPIK-P1 data cut-off date) to the day before the first interventional dose of alpelisib is administered in the prospective period of this study (Day -1). Prospective: From Day 1 up to 5 years
  Proportion of participants requiring PROS-related treatment(s) other than alpelisib, including medications (concomitant PROS-related medications including medication for the management of PROS related complications as well as medications to manage complications secondary to alpelisib) and non-drug treatments (e.g., feeding tube, ketogenic diet, non-invasive device for sleep apnea, sclerotherapy, endovascular occlusive procedures)
Retrospective and prospective period: Proportion of participants with dose adjustments of alpelisib | Retrospective: From 10-Mar-2020 (1 day after EPIK-P1 data cut-off date) to the day before the first interventional dose of alpelisib is administered in the prospective period of this study (Day -1). Prospective: From Day 1 up to 5 years
  Proportion of participants requiring dose increase, reductions and interruptions of alpelisib
Retrospective and prospective period: Proportion of participants with PROS-related surgeries | Retrospective: From 10-Mar-2020 (1 day after EPIK-P1 data cut-off date) to the day before the first interventional dose of alpelisib is administered in the prospective period of this study (Day -1). Prospective: From Day 1 up to 5 years
  Proportion of participants requiring surgery due to PROS

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- Boston Childrens Hospital, Boston, Massachusetts, United States
- France (3):
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
- Novartis Investigative Site, Dublin, Ireland
- Novartis Investigative Site, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com